CLINICAL TRIAL: NCT04293575
Title: MitraBridge Registry
Brief Title: Transcatheter Mitral Valve Repair as Bridge Therapy to Heart Transplantation
Acronym: MitraBridge
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Cosmo Godino, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: MITRABRIDGE280220
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Mitral Regurgitation; End-stage Heart Failure
Keywords: transcatheter mitral valve repair; mitraclip; heart transplantation; LVAD
MeSH Terms: conditions — Heart Failure; Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- In list group: patients on active heart transplantation (HTx) list with a low likelihood to receive a donation shortly (e.g. for body weight or blood group)
  Interventions: Device: MitraClip
- Bridge to decision "BTD" group: patients suitable for HTx, but that were still waiting for clinical decision
  Interventions: Device: MitraClip
- (Bridge to candidacy "BTC" group): patients who could not be yet in list for HTx because of concomitant, potentially reversible, contraindications such as severe pulmonary hypertension, elevated pulmonary-vascular-resistance, unsatisfactory response to vasodilator challenge or other causes resulting in a prohibitive peri-procedural risk (as pre-transplant body mass index [BMI] >35 kg/m2, severe renal dysfunction with creatinine clearance <30 mL/min) and other reasons (current alcohol, tobacco or drug abuse, poor social support, non-residents)
  Interventions: Device: MitraClip

INTERVENTIONS:
Device: MitraClip — transcatheter MitraClip device (Abbott Vascular, Santa Clara, California)

SUMMARY:
The aim of this study is to report medium-term outcomes after the use of transcatheter mitral valve repair (TMVR) with MitraClip as a bridge therapy to heart transplantation (HTx) in patients with mitral regurgitation (MR) and end-stage heart failure (HF).

DETAILED DESCRIPTION:
Background: Heart transplantation (HTx) is the most effective therapeutic option for patients with advanced or end-stage chronic heart failure (HF). However, the increasing number of patients with refractory chronic HF and the declining willingness for organ donation, have resulted in expanded waiting lists and prolonged waiting times for patients listed for HTx. Furthermore, more than 60% of patients are transplanted in high-urgency status, leaving little chance for patients listed for less urgent transplantation. In order to improve the general conditions of these latter patients during the waiting period, several pharmacological and mechanical bridging therapies have been developed. Anyway, limited data are now available regarding the use of MitraClip treatment as bridge strategy in patients with severe mitral regurgitation (MR) and end-stage HF waiting for HTx.

Methods: The MitraBridge registry is an observational, multicenter, international registry including all consecutive patients with chronic end-stage HF [New York Heart Association (NYHA) III or IV and/or left ventricular ejection fraction (LVEF) ≤35%] and concomitant moderate-severe or severe MR who were potential candidates for HTx, that were treated with MitraClip in the contest of a pre-specified bridge strategy.

According to the clinical conditions present at the time of the MitraClip procedure, patients are classified in:

1. patients on active HTx list (In list group, "pure bridge") with a rapidly progressive disease and a low likelihood to receive a donation shortly;
2. patients waiting for clinical decision (Bridge to decision "BTD" group), also including unstable patients during the screening for HTx;
3. patients who could not be listed for HTx (Not in list group, MitraClip as "bridge to candidacy") because of concomitant, potentially reversible, contraindications (e.g. severe pulmonary hypertension, elevated pulmonary-vascular-resistance).

The registry was initiated in June 2018 without the support of any external funding and was designed to involve centers across the world that have experience with transcatheter MitraClip device (Abbott Vascular, Santa Clara, California).

Study endpoints. The primary endpoint: 1-year composite adverse events rate of all-cause of death, urgent/unplanned HTx or LVAD implantation and first re-hospitalization for HF.

As exploratory outcomes: individual components of the primary endpoint.

Moreover, the investigators described the clinical status of patients at the time of last available follow-up, in order to report the rates of patients going for elective HTx, entering (or remaining) in the waiting list and having no more indication to HTx (delisting) because of significant echocardiographic and/or clinical improvements during the entire observational period.

Mitral Valve Academic Research Consortium (MVARC) criteria are used to define procedural success and composite events 12.

Follow-up data will be collected for patients at 1 month and 1-year and then according to the time frame elapsed from the index procedure to data lock for present analysis.

Patients that did not implant any clip during the index procedure were not included in the follow-up. For patients who underwent HTx or LVAD implantation, the follow-up time was stopped at the date of transplant or mechanical device placement.

ELIGIBILITY:
Inclusion Criteria:

* patients with chronic end-stage HF [New York Heart Association (NYHA) III or IV and/or left ventricular ejection fraction (LVEF) ≤35%] and concomitant moderate-severe or severe MR being potential candidates for HTx.
* patients on active HTx list (In list group, "pure bridge") with a low likelihood to receive a donation shortly (e.g. for body weight or blood group);
* patients suitable for HTx, but that were still waiting for clinical decision (Bridge to decision, "BTD" group);
* patients who could not be yet in list for HTx (Bridge to candidacy, "BTC" group) because of concomitant, potentially reversible, contraindications such as severe pulmonary hypertension, elevated pulmonary-vascular-resistance, unsatisfactory response to vasodilator challenge or other causes resulting in a prohibitive peri-procedural risk (as pre-transplant body mass index [BMI] >35 kg/m2, severe renal dysfunction with creatinine clearance <30 mL/min) and other reasons (current alcohol, tobacco or drug abuse, poor social support, non-residents)

Exclusion Criteria:

* patients with mitral valve anatomy not suitable for percutaneous mitral valve repair using the MitraClip device

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All potential candidates for HTx treated with MitraClip in the contest of a pre-specified bridge strategy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite adverse events rate of all-cause of death, urgent/unplanned HTx or LVAD implantation and first re-hospitalization for HF | up to 1-year since the MitraClip procedure
  1-year Rate of composite adverse events of all-cause of death, urgent/unplanned HTx or LVAD implantation and first re-hospitalization for HF

SECONDARY OUTCOMES:
All-cause of death | up to 1-year since the MitraClip procedure
  Rate of all-cause of death
Urgent/unplanned HTx | up to 1-year since the MitraClip procedure
  Rate of urgent/unplanned HTx
Urgent/unplanned LVAD | up to 1-year since the MitraClip procedure
  Rate of urgent/unplanned LVAD
First re-hospitalization for HF | up to 1-year since the MitraClip procedure
  Rate of first re-hospitalization for HF

OTHER OUTCOMES:
Rate of patients going for elective HTx, entering (or remaining) in the waiting list and having no more indication to HTx (delisting) because of significant echocardiographic and/or clinical improvements during the entire observational period. | up to 1-year since the MitraClip procedure
  Rate of patients going for elective HTx, entering (or remaining) in the waiting list and no more indication to HTx (delisting) because of significant echocardiographic and/or clinical improvements during the entire observational period.

CONTACTS AND LOCATIONS:
Locations (1):
- Cosmo Godino, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months